CLINICAL TRIAL: NCT03667729
Title: The Effects of Progressive Muscle Relaxation Therapy in Patients With Schizophrenia: Randomized Controlled Trials
Brief Title: The Effects of Progressive Muscle Relaxation Therapy in Patients With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: C20140205
Record Dates: First submitted 2018-08-20; First posted 2018-09-12 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2017-06

CONDITIONS: Affective Disorders; Psychotic Disorder
Keywords: PMR, anxiety, psychotic syndrome, quality of life
MeSH Terms: conditions — Mood Disorders; Psychotic Disorders; Anxiety Disorders | interventions — Autogenic Training

STUDY DESIGN:
Intervention Model Description: This study applied a randomized parallel case-controlled design.
  Hospital-based randomized control trial . Subjects were chronic schizophrenia who were recruited from a psychotic ward complex and randomized into PMR, or control groups.
Who Masked: Outcomes Assessor
Masking Description: The rater did not know what interventions the participants belonged to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- progressive muscle relaxation (Experimental): The experimental group received PMR once a week for a total of 12 weeks. Subjects completed measures at baseline, 3-month, and 3-month follow-up.
  Interventions: Behavioral: progressive muscle relaxation
- Control group (No Intervention): treatment-as-usual(TAU)

INTERVENTIONS:
Behavioral: progressive muscle relaxation — intervention group: The experimental group received muscle relaxation training once a week for 3 consecutive months. The results were measured and followed up after 3 months.
  Arms: progressive muscle relaxation

SUMMARY:
This study applied a randomized parallel case-controlled design. The study purpose was to evaluate the effects of progressive muscle relaxation on anxiety, psychiatric symptoms and quality of life among patients with chronic schizophrenia compared with an active control.

DETAILED DESCRIPTION:
Background: Anti-psychotic drugs are limited in their ability to improve psychiatric symptoms, quality of life, and anxiety status in patients with chronic schizophrenia. Progressive Muscle Relaxation (PMR) can potentially reduce anxiety status and improve subjective welling in acute patients. It is an ideal rehabilitation intervention for patients with chronic schizophrenia. However, no study has investigated the effects of PMR on outcomes among patients with chronic schizophrenia.

Design: This study applied a randomized parallel case-controlled design.

Methods: Hospital-based randomized control trial in Taiwan. Eighty subjects with chronic schizophrenia were recruited from a psychotic ward and randomized into PMR, or control groups. Patients in the intervention group participated in progressive muscle relaxation for 12 weeks; while patients in the control group members received supportive treatment-as-usual (TAU). All participants completed anxiety, psychotic syndromes and quality of life measures at baseline, 3-month, and 3-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Schizophrenia
* Without the risk of self-injury and violence
* Patients aged from 20-65 years old
* Had no alcohol and drug abuse
* Can use Mandarin or Taiwanese to communicate

Exclusion Criteria:

* Patients with another psychiatric comorbidity
* Patients with musculoskeletal problems
* patients who cannot sit last for 50 minutes
* Had received progressive muscle relaxation training within the last year
* Diagnosis of confirmed cardiovascular disease

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2014-06-30 (Actual); Primary Completion 2015-06-29 (Actual); Study Completion 2015-06-29 (Actual)

PRIMARY OUTCOMES:
Quality of life simplified Chinese versions of the WHOQOL-BREF questionnaire were used | Measuring changes in quality of life from baseline to 6 months.
  a 28-item questionnaire rated on a five-point Likert scale with four domains measuring: psychological health, physical health, social relationships and environment.so that higher scores refer to high QOL.

SECONDARY OUTCOMES:
Anxiety Scale | measured at baseline, 3-month, and 3-month follow-up
  State anxiety was assessed by the State anxiety inventory (SAI) of Spielberg (1984). The range of possible total scores is 20-80. Higher scores indicate higher levels of anxiety.
Positive and Negative Syndrome Scale (PANSS) | measured at baseline, 3-month, and 3-month follow-up
  The instrument was developed by Kay et al. (1987) to assess psychopathology of schizophrenia which includes: positive, negative, general psychopathology symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: hsiu-ju Chang, PHD, Principal Investigator — Taipei Medical University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bernstein, D. A., & Borkovec, T. D. (1973). Progressive Relaxation Training: A Manual for the Helping Professions.
- [Background] SpielBerger C. (1983). Manual for the state-trait anxiety inventory. Palo Alto, CA: Consulting Psychologists Press.
- [Background] Hedlund, J. L. & Vieweg, B. W. (1980) The Brief Psychiatric Rating Scale (BPRS): a comprehensive review. Journal of Operational Psychiatry, 11, 48- 65.
- [Background] Bernstein, D. & Borkove, c. T. (1973). Progressive relaxation training. Champaign, IL: Research Press.
- [Background] Overall, J.E., Gorham, D.R., 1962. The brief psychiatric rating scale. Psychol. Rep. 10, 799e812.
- [Background] Overall, J.E., 1974. The brief psychiatric rating scale in psychopharmacology research. In: Pichot, P., Olivier-Martin, E. (Eds.), Psychological Measurements in Psychopharmacology: Modern Problems in Psychopharmacology. Karger, Basel, Switzerland, pp. 67e78.
- [Result] Ben-Zeev D, Larson J, Sarratt M. A possible role for Progressive Muscle Relaxation in the treatment of persecutory ideation. Med Hypotheses. 2010 Dec;75(6):568-71. doi: 10.1016/j.mehy.2010.07.033. Epub 2010 Aug 14. PMID 20709459
- [Result] Bebbington PE, Angermeyer M, Azorin JM, Marwaha S, Marteau F, Toumi M. Side-effects of antipsychotic medication and health-related quality of life in schizophrenia. Acta Psychiatr Scand Suppl. 2009;(438):22-8. doi: 10.1111/j.1600-0447.2008.01310.x. PMID 19132963
- [Result] Achalia RM, Chaturvedi SK, Desai G, Rao GN, Prakash O. Prevalence and risk factors associated with tardive dyskinesia among Indian patients with schizophrenia. Asian J Psychiatr. 2014 Jun;9:31-5. doi: 10.1016/j.ajp.2013.12.010. Epub 2014 Jan 4. PMID 24813033
- [Result] Chino B, Nemoto T, Fujii C, Mizuno M. Subjective assessments of the quality of life, well-being and self-efficacy in patients with schizophrenia. Psychiatry Clin Neurosci. 2009 Aug;63(4):521-8. doi: 10.1111/j.1440-1819.2009.01995.x. Epub 2009 Jun 15. PMID 19531107
- [Result] Cramer H, Lauche R, Klose P, Langhorst J, Dobos G. Yoga for schizophrenia: a systematic review and meta-analysis. BMC Psychiatry. 2013 Jan 18;13:32. doi: 10.1186/1471-244X-13-32. PMID 23327116
- [Result] Erol A, Delibas H, Bora O, Mete L. The impact of insight on social functioning in patients with schizophrenia. Int J Soc Psychiatry. 2015 Jun;61(4):379-85. doi: 10.1177/0020764014548287. Epub 2014 Sep 1. PMID 25182810
- [Result] Georgiev A, Probst M, De Hert M, Genova V, Tonkova A, Vancampfort D. Acute effects of progressive muscle relaxation on state anxiety and subjective well-being in chronic Bulgarian patients with schizophrenia. Psychiatr Danub. 2012 Dec;24(4):367-72. PMID 23132187
- [Result] Hartley S, Barrowclough C, Haddock G. Anxiety and depression in psychosis: a systematic review of associations with positive psychotic symptoms. Acta Psychiatr Scand. 2013 Nov;128(5):327-46. doi: 10.1111/acps.12080. Epub 2013 Feb 4. PMID 23379898
- [Result] Harvey PD, Loewenstein DA, Czaja SJ. Hospitalization and psychosis: influences on the course of cognition and everyday functioning in people with schizophrenia. Neurobiol Dis. 2013 May;53:18-25. doi: 10.1016/j.nbd.2012.10.022. Epub 2012 Oct 31. PMID 23123218
- [Result] Holubova M, Prasko J, Hruby R, Latalova K, Kamaradova D, Marackova M, Slepecky M, Gubova T. Coping strategies and self-stigma in patients with schizophrenia-spectrum disorders. Patient Prefer Adherence. 2016 Jun 24;10:1151-8. doi: 10.2147/PPA.S106437. eCollection 2016. PMID 27445463
- [Result] Hunter R, Barry S. Negative symptoms and psychosocial functioning in schizophrenia: neglected but important targets for treatment. Eur Psychiatry. 2012 Aug;27(6):432-6. doi: 10.1016/j.eurpsy.2011.02.015. Epub 2011 May 23. PMID 21602034
- [Result] Jeyagurunathan A, Vaingankar JA, Abdin E, Sambasivam R, Seow E, Pang S, Picco L, Chong SA, Subramaniam M. Gender differences in positive mental health among individuals with schizophrenia. Compr Psychiatry. 2017 Apr;74:88-95. doi: 10.1016/j.comppsych.2017.01.005. Epub 2017 Jan 12. PMID 28113098
- [Result] Karow A, Wittmann L, Schottle D, Schafer I, Lambert M. The assessment of quality of life in clinical practice in patients with schizophrenia. Dialogues Clin Neurosci. 2014 Jun;16(2):185-95. doi: 10.31887/DCNS.2014.16.2/akarow. PMID 25152657
- [Result] Karpov B, Joffe G, Aaltonen K, Suvisaari J, Baryshnikov I, Naatanen P, Koivisto M, Melartin T, Oksanen J, Suominen K, Heikkinen M, Paunio T, Isometsa E. Anxiety symptoms in a major mood and schizophrenia spectrum disorders. Eur Psychiatry. 2016 Sep;37:1-7. doi: 10.1016/j.eurpsy.2016.04.007. Epub 2016 Jul 21. PMID 27447101
- [Result] Kay SR, Fiszbein A, Opler LA. The positive and negative syndrome scale (PANSS) for schizophrenia. Schizophr Bull. 1987;13(2):261-76. doi: 10.1093/schbul/13.2.261. PMID 3616518
- [Result] Lecardeur L. [The quality of life in schizophrenia]. Encephale. 2015 Sep;41(4):373-8. doi: 10.1016/j.encep.2015.07.001. Epub 2015 Sep 2. French. PMID 26341538
- [Result] Li Y, Hou CL, Ma XR, Zhong BL, Zang Y, Jia FJ, Lin YQ, Lai KYC, Chiu HFK, Ungvari GS, Hall BJ, Cai MY, Ng CH, Xiang YT. Quality of life in Chinese patients with schizophrenia treated in primary care. Psychiatry Res. 2017 Aug;254:80-84. doi: 10.1016/j.psychres.2017.04.049. Epub 2017 Apr 24. PMID 28456026
- [Result] Marder SR, Galderisi S. The current conceptualization of negative symptoms in schizophrenia. World Psychiatry. 2017 Feb;16(1):14-24. doi: 10.1002/wps.20385. PMID 28127915
- [Result] Margariti M, Ploumpidis D, Economou M, Christodoulou GN, Papadimitriou GN. Quality of life in schizophrenia spectrum disorders: associations with insight and psychopathology. Psychiatry Res. 2015 Feb 28;225(3):695-701. doi: 10.1016/j.psychres.2014.11.016. Epub 2014 Nov 15. PMID 25544550
- [Result] Mas-Exposito L, Amador-Campos JA, Gomez-Benito J, Lalucat-Jo L. The World Health Organization Short Disability Assessment Schedule: a validation study in patients with schizophrenia. Compr Psychiatry. 2012 Feb;53(2):208-16. doi: 10.1016/j.comppsych.2011.02.009. Epub 2011 Apr 12. PMID 21489417
- [Result] McGrath J, Saha S, Chant D, Welham J. Schizophrenia: a concise overview of incidence, prevalence, and mortality. Epidemiol Rev. 2008;30:67-76. doi: 10.1093/epirev/mxn001. Epub 2008 May 14. PMID 18480098
- [Result] Mingrone C, Rocca P, Castagna F, Montemagni C, Sigaudo M, Scalese M, Rocca G, Bogetto F. Insight in stable schizophrenia: relations with psychopathology and cognition. Compr Psychiatry. 2013 Jul;54(5):484-92. doi: 10.1016/j.comppsych.2012.12.014. Epub 2013 Jan 15. PMID 23332554
- [Result] Muller DJ, Chowdhury NI, Zai CC. The pharmacogenetics of antipsychotic-induced adverse events. Curr Opin Psychiatry. 2013 Mar;26(2):144-50. doi: 10.1097/YCO.0b013e32835dc9da. PMID 23370274
- [Result] Oliveira SE, Carvalho H, Esteves F. Toward an understanding of the quality of life construct: Validity and reliability of the WHOQOL-Bref in a psychiatric sample. Psychiatry Res. 2016 Oct 30;244:37-44. doi: 10.1016/j.psychres.2016.07.007. Epub 2016 Jul 8. PMID 27455149
- [Result] Pallanti S, Quercioli L, Hollander E. Social anxiety in outpatients with schizophrenia: a relevant cause of disability. Am J Psychiatry. 2004 Jan;161(1):53-8. doi: 10.1176/appi.ajp.161.1.53. PMID 14702250
- [Result] Pelka M, Kolling S, Ferrauti A, Meyer T, Pfeiffer M, Kellmann M. Acute effects of psychological relaxation techniques between two physical tasks. J Sports Sci. 2017 Feb;35(3):216-223. doi: 10.1080/02640414.2016.1161208. Epub 2016 Mar 21. PMID 26999625
- [Result] Rofail D, Regnault A, le Scouiller S, Berardo CG, Umbricht D, Fitzpatrick R. Health-related quality of life in patients with prominent negative symptoms: results from a multicenter randomized Phase II trial on bitopertin. Qual Life Res. 2016 Jan;25(1):201-11. doi: 10.1007/s11136-015-1057-9. Epub 2015 Jul 5. PMID 26143058
- [Result] Tandon R, Gaebel W, Barch DM, Bustillo J, Gur RE, Heckers S, Malaspina D, Owen MJ, Schultz S, Tsuang M, Van Os J, Carpenter W. Definition and description of schizophrenia in the DSM-5. Schizophr Res. 2013 Oct;150(1):3-10. doi: 10.1016/j.schres.2013.05.028. Epub 2013 Jun 22. PMID 23800613
- [Result] Tsou JY. Natural kinds, psychiatric classification and the history of the DSM. Hist Psychiatry. 2016 Dec;27(4):406-424. doi: 10.1177/0957154X16656580. Epub 2016 Jul 4. PMID 27378802
- [Result] Vancampfort D, Correll CU, Scheewe TW, Probst M, De Herdt A, Knapen J, De Hert M. Progressive muscle relaxation in persons with schizophrenia: a systematic review of randomized controlled trials. Clin Rehabil. 2013 Apr;27(4):291-8. doi: 10.1177/0269215512455531. Epub 2012 Jul 27. PMID 22843353
- [Result] Vancampfort D, De Hert M, Knapen J, Maurissen K, Raepsaet J, Deckx S, Remans S, Probst M. Effects of progressive muscle relaxation on state anxiety and subjective well-being in people with schizophrenia: a randomized controlled trial. Clin Rehabil. 2011 Jun;25(6):567-75. doi: 10.1177/0269215510395633. Epub 2011 Mar 14. PMID 21402653
- [Result] Vancampfort D, De Hert M, Knapen J, Wampers M, Demunter H, Deckx S, Maurissen K, Probst M. State anxiety, psychological stress and positive well-being responses to yoga and aerobic exercise in people with schizophrenia: a pilot study. Disabil Rehabil. 2011;33(8):684-9. doi: 10.3109/09638288.2010.509458. Epub 2010 Aug 18. PMID 20718623
- [Result] Vancampfort D, Probst M, Helvik Skjaerven L, Catalan-Matamoros D, Lundvik-Gyllensten A, Gomez-Conesa A, Ijntema R, De Hert M. Systematic review of the benefits of physical therapy within a multidisciplinary care approach for people with schizophrenia. Phys Ther. 2012 Jan;92(1):11-23. doi: 10.2522/ptj.20110218. Epub 2011 Nov 3. PMID 22052946
- [Result] Vera-Garcia E, Mayoral-Cleries F, Vancampfort D, Stubbs B, Cuesta-Vargas AI. A systematic review of the benefits of physical therapy within a multidisciplinary care approach for people with schizophrenia: An update. Psychiatry Res. 2015 Oct 30;229(3):828-39. doi: 10.1016/j.psychres.2015.07.083. Epub 2015 Jul 31. PMID 26254795
- [Result] Wang FZ, Luo D, Kanb W, Wang Y. Combined intervention with education and progressive muscle relaxation on quality of life, functional disability, and positive symptoms in patients with acute schizophrenia. J Altern Complement Med. 2015 Mar;21(3):159-65. doi: 10.1089/acm.2014.0128. Epub 2015 Feb 11. PMID 25671655
- [Result] The World Health Organization Quality of Life assessment (WHOQOL): position paper from the World Health Organization. Soc Sci Med. 1995 Nov;41(10):1403-9. doi: 10.1016/0277-9536(95)00112-k. PMID 8560308